CLINICAL TRIAL: NCT03281421
Title: Immediate Effects of Ankle Mobilization on Dorsiflexion Range of Motion in Closed Kinetic Chain in Women With Patellofemoral Pain: A Random Clinical Trial
Brief Title: Immediate Effects of Ankle Mobilization on Dorsiflexion Range of Motion in Women With Patellofemoral Pain.
Acronym: Mestrado
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Gabriel Peixoto Leão Almeida, Professor, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mestrado_Bruno
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group from posterior to anterior (GPA) (Experimental): Participants in group GPA will receive a manual therapy intervention, through the technique of mobilization with movement in the ankle joint, with a slip sense from posterior to anterior. The physiotherapist will be positioned in front the participant's ankle, and a belt will be posicioned above the participant's malleolus and around physiotherapist's pelvis. The therapist applies with belt a anterior slip sustained in the tibia of the participant, while the talus are secured with the space between the thumb and the second finger of the hand of both hands on the physiotherapist´s. The participant will be instructed to perform a slow dorsiflexion movement at its maximum amplitude and hold five seconds in that position, returning to the initial position at the end of the five seconds.
  Interventions: Other: Manual Therapy
- Group from anterior to posterior (GAP) (Active Comparator): Participants in group GAP will receive a manual therapy intervention, through the technique of mobilization with movement in the ankle joint, with a slip sense from anterior to posterior. The physiotherapist will be positioned behind the participant's ankle. An belt will be posicioned above the participant's malleolus and around physiotherapist's trunk. The therapist applies with belt a posterior slip sustained in the tibia of the participant, while the heel and rearfoot are secured with the space between the thumb and the second finger of the hand of both hands on the physiotherapist´s. The participant will be instructed to perform a slow dorsiflexion movement at its maximum amplitude and hold five seconds in that position, returning to the initial position at the end of the five seconds.
  Interventions: Other: Manual Therapy
- Group GPA-AP (Active Comparator): Participants in group GAP will receive a manual therapy intervention, through the technique of mobilization with movement in the ankle joint, with a slip sense both from posterior to anterior and anterior to posterior. In the group GPA-AP, will be apllied both the procedure described for the group GPA as for the group GAP. To standardized the sequence of mobilization, the first two sets will be performed with slip sense from posterior to anterior, and the last two sets will be performede with slip sense from anterior to posterior.
  Interventions: Other: Manual Therapy

INTERVENTIONS:
Other: Manual Therapy — The manual therapy intervention, through the technique of mobilization with movement in the ankle joint (following the specific sense direction of the group), will be performed in a protocol that consists of four sets of five repetitions, with rest time between series of one minute.
  Other Names: Manual Physical Therapy

SUMMARY:
Anterior Knee Pain or Patellofemoral Pain (PFP) is one of the most common disorders that affecting knee in the physically active population, being a condition that typically presents as diffuse knee pain in the anterior region and retro- or peri-patellar area, mainly in activities that increase compression force in patellofemoral joint, such as squatting, running, stair ascent and descent. The overall prevalence of PFP has been reported as between 15-45% of the population, and its incidence is higher among women. The literature cites as etiology of PFP the ocorrence of dysfunctions in the local (knee), proximal (trunk, pelvis and hip complex) and distal (ankle and foot regions) factores. Actually, there is a lack of studies that investigate the interventions influences on distal factors in outcomes clinical in persons with PFP. Thus, the aim of this study is analyze the effect of ankle mobilization techiniques in ankle dorsiflexion range of motion closed kinetic chain in women with patellofemoral pain and with dorsoflexion restriction.

DETAILED DESCRIPTION:
The sample of this study will be formed by 117 lower limbs of women with PFP who have ankle dorsoflexion restriction, divided into three groups. Each group will contain 39 lower limbs and receive an ankle mobilization technique with a specific sense of mobilization. The group nominated GAP will receive an mobilization technique with slip sense from anterior to posterior. The group nominated GPA will receive an mobilization technique with slip sense from posterior to anterior. The group nominated GPA-AP will receive an mobilization technique with slip sense both from posterior to anterior and from anterior to posterior.

Each group will receive a single intervention, which will consist of four sets of five repetitions of the ankle mobilization technique (according to the specific slip direction of each group), with rest time between series of one minute. In the group GPA-AP, to standardized the sequence of mobilization, the first two sets will be performed with slip sense from anterior to posterior, and the last two sets will be performede with slip sense from posterior to anterior. There will be randomisation allocation of individuals in the groups and because of the nature of the interventions only the evaluator may be blind.

The Kolmogorov - Smirnov test is used to verify the data distribution normality. The characterization of the participants is performed by means of descriptive statistical analysis. Parametric or non-parametric tests will be used according to the data distribution normality for comparison between groups at baseline. The evaluator blinding will be tested using the chi -square test by comparing the randomization code with the evaluator opinion. The difference between the groups and their respective confidence intervals will be calculated by linear mixed models using interaction term of "time versus group".

ELIGIBILITY:
Inclusion Criteria:

* Presence of localized pain in the anterior region of the knee and / or around the patella, reproduced with at least two of the following activities: climbing / descending stairs, crouching, kneeling, long sitting, isometric contraction of the quadriceps, running and jump.
* Existence of a report of pain for at least three months, beginning incidental and unrelated to some traumatic event in the knee.
* Pain with intensity of at least three points in the Visual Analogue Scale (VAS) of pain in the last week.
* Limitation of the ankle dorsiflexion range of motion measured by the Lunge Test in the lower limb with Patellofemoral Pain.

Exclusion Criteria:

* History of surgery in the lumbar spine, hip, knee and / or ankle;
* History of fractures in the lumbar spine, hip, knee and / or ankle;
* History of patellar dislocation;
* Presence of edema in the knee joint;
* Presence of meniscal injury;
* Injury of cruciate ligament and / or collateral ligaments;
* Presence of tendonopathy in the patellar tendon, tendons of the goose and / or band leg tibial ilium;
* Presence of Osgood-Schlatter Syndrome or Sinding-Larsen-Johansson Syndromes.
* Presence of pain in the lumbar spine and / or hip.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Range of motion of ankle dorsiflexion. | Immediatly after intervention day.
  Closed kinetic chain evaluation to find the greatest distance between the foot and the wall without compensations.

SECONDARY OUTCOMES:
Range of motion of ankle dorsiflexion. | Two days after intervention day.
  Closed kinetic chain evaluation to find the greatest distance between the foot and the wall without compensations.
Angle of projection in the frontal plane in the lower limb. | Immediatly and two days after intervention day.
  Will be measured during the conduct of the Forward Step-Down Test through captured footage using a digital camera that will be positioned within two meters of the participant.
Numeric Pain Scale. | Immediatly and two days after intervention day.
  Pain was assessed by use of an Numeric Pain Scale of eleven point, where zero corresponded to no pain and ten corresponded to worst imaginable pain
Global Effect Perception Scale for Treatment | Immediatly and two days after intervention day.
  Global Effect Perception Scale for Treatment was assessed by use f an numeric scale of eleven point, where the lowest score corresponds to the extremely worst condition and the highest score corresponds to the fully recovered condition.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel PL Almeida, MSc, Principal Investigator — Federal University of Ceará (UFC), Brazil.
Locations (1):
- Federal University of Ceara, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No